CLINICAL TRIAL: NCT00950508
Title: European Multicenter Plasma Exchange Trial (Empet): A Controlled, Open, Randomised, Multicenter Study In Patients With Acute Liver Failure
Brief Title: A Study of the Effect of Plasmaexchange in Patients With Acute Liver Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Dr. Fin Stolze Larsen, Senior consultant, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMPET-001
Record Dates: First submitted 2009-07-29; First posted 2009-07-31 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Acute Liver Failure
MeSH Terms: conditions — Liver Failure, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High volume plasma exchange (Active Comparator): 3 successive plasma exchanges over 3 days
  Interventions: Procedure: High volume plasma exchange; Procedure: Standard medical treatment
- Standard medical treatment (Placebo Comparator)
  Interventions: Procedure: Standard medical treatment

INTERVENTIONS:
Procedure: High volume plasma exchange — 3 high volume plasma exchanges over 3 days
  Other Names: HVP
  Arms: High volume plasma exchange
Procedure: Standard medical treatment — Standard medical treatment
  Other Names: SMT

SUMMARY:
The aim of this study is to examine if high-volume plasma exchange has a positive effect on mortality in patients with acute liver failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute liver failure in encephalopathy grade 2-4

Exclusion Criteria:

* alcoholic hepatitis
* primary non function liver graft or graft dysfunction
* known chronic liver disease
* known malignancies
* clinical suspicion of brain death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 1998-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
mortality | at day 3, day 7

CONTACTS AND LOCATIONS:
Overall Officials: Fin S Larsen, PhD,Dr.M.Sc, Study Chair — Rigshospitalet, Denmark
Locations (3):
- Department of Hepatology, Rigshospitalet, Copenhagen, DK, Denmark
- Department of Transplantation and Liver Surgery, Helsinki University Hospital, Helsinki, Finland
- Institute of Liver Studies, King's College Hospital, London, United Kingdom

REFERENCES:
- [Derived] Larsen FS, Schmidt LE, Bernsmeier C, Rasmussen A, Isoniemi H, Patel VC, Triantafyllou E, Bernal W, Auzinger G, Shawcross D, Eefsen M, Bjerring PN, Clemmesen JO, Hockerstedt K, Frederiksen HJ, Hansen BA, Antoniades CG, Wendon J. High-volume plasma exchange in patients with acute liver failure: An open randomised controlled trial. J Hepatol. 2016 Jan;64(1):69-78. doi: 10.1016/j.jhep.2015.08.018. Epub 2015 Aug 29. PMID 26325537